CLINICAL TRIAL: NCT05921669
Title: The Effect Of Traınıng On Breastfeedıng Gıven To Fathers On Breastfeedıng, Parent-Baby Bondıng And Breastfeedıng Self-Effıcacy Level
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, İLFAN KARANFİL, Nurse, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: EskisehirOU-IKARANFIL-001-001
Record Dates: First submitted 2023-03-26; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Breast Feeding
Keywords: breastfeeding; paternal support; child health
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Before starting the research, parents will be informed about the study and written consent will be obtained from those who agree to participate in the research. There are 3 groups in the study. These; Experimental Group 1: The group in which breastfeeding training was given to mothers and fathers Experimental Group 2: The group in which breastfeeding training was given only to the mother Control Group: The group that did not receive any intervention and received routine hospital care.
  Within the first 24 hours after birth, everyone participating in the research will be contacted and the relevant forms will be filled in and breastfeeding training will be given to experimental group 1 and experimental group 2 by the researcher. Then, families will be called in the 1st week, 1st month and 3rd month by phone and the relevant forms will be filled. Families' questions about breastfeeding will be answered.
Who Masked: Participant, Outcomes Assessor
Masking Description: The lottery method and blocking will be used in assigning individuals to groups. Participants will be laided according to the way of birth and then the draw will be divided into groups. For the first person to be included in the study in the lottery method; In a bag of the same size and the same quality, three separate paper on which "Control Group", "Mother Training Group", "Mother and Father Education Group" will be placed. The first participant will be determined in this way. For the second participant; 2 paper containing groups not including the first participant will be thrown into the bag and draw the draw. In the third participant, the draw will not be drawn, and the person will be appointed to the remaining group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group 1: The group in which breastfeeding training was given to mothers and fathers (Experimental): Face-to-face theoretical breastfeeding training and then practical training (breastfeeding techniques, burping, changing diapers, milking by hand or pump, etc.) will be given by the researcher to the mothers and fathers. This training is planned to take 30-45 minutes. Then, an additional 15-30 minutes of father-supported breastfeeding training will be given to fathers. At the end of the training, the "Breastfeeding Booklet" prepared by the researchers will be given to the parents.
  Interventions: Behavioral: Provide breastfeeding education
- Experimental Group 2: The group in which breastfeeding training was given only to the mother (Experimental): Only mothers will receive face-to-face theoretical breastfeeding training followed by practical training (breastfeeding techniques, flatulence, changing diapers, milking by hand or pump, etc.). This training is planned to take 30-45 minutes. At the end of the training, mothers will be given a "Breastfeeding Booklet" prepared by the researchers.
  Interventions: Behavioral: Provide breastfeeding education
- Control Group: No intervention was made, group receiving routine hospital care) (No Intervention): No additional training will be given to this group by the researcher, apart from the trainings included in the routine procedures of the hospital.

INTERVENTIONS:
Behavioral: Provide breastfeeding education — Providing breastfeeding education within the first 24 hours after birth
  Arms: Experimental Group 1: The group in which breastfeeding training was given to mothers and fathers; Experimental Group 2: The group in which breastfeeding training was given only to the mother

SUMMARY:
The most suitable food for babies is breast milk. It is known that breastfeeding, beyond providing nutrition, has many health benefits for the baby and the mother. The World Health Organization (WHO) recommends that babies start breastfeeding within 1 hour after birth and breastfeed exclusively without any additional food, including water, for the first 6 months. After six months, complementary foods should be started, and the baby should continue to be breastfed for two years or more. On the other hand, between 2015-2020, the rates of infants aged 0-6 months fed with breast milk alone are approximately 44% worldwide.

There are many factors that affect the time of initiation of breastfeeding and the duration of breastfeeding. Some of those; maternal education, mode of delivery, birth weight and socio-economic status. Another influential factor is paternal support. Fathers may want to be involved in breastfeeding education and support their spouses in this process. However, the reasons such as not taking part in the trainings and not being asked direct questions about breastfeeding may cause fathers to feel excluded in this process. It is important to include fathers in education and interventions to achieve breastfeeding goals. Mothers who are supported by their spouses during the breastfeeding process experience breastfeeding problems less and can cope with these problems better.

Today, it is known that fathers are not given sufficient importance in promoting breastfeeding. Including fathers in breastfeeding education can increase the rate and duration of breastfeeding of infants. This study was planned to determine the effect of breastfeeding education given to mothers and/or fathers in the postnatal period on breastfeeding, parent-infant attachment and breastfeeding self-efficacy. The aim of the study is to draw attention to the importance of father support in breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

* Parent's consent to participate in the research
* Parents must be at least primary school graduates
* Mothers and fathers to participate in the study must be 20 years or older
* The mother's first pregnancy (primiparous pregnant)
* Having a smart mobile phone of the mother and father
* The baby is born at term

Exclusion Criteria:

* Experiencing communication problems with parents (mother and father cannot speak and/or understand Turkish, etc.)
* Having or developing a health problem in the mother or baby
* Separation of the mother from her baby for any reason after birth

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Breastfeeding Self-Efficacy Scale-short form | 3 months
  The short version of the breastfeeding self-efficacy scale consisted of a total of 14 items evaluating breastfeeding self-efficacy. The scale is in a 5-point Likert type and is evaluated as 1 = I am not sure at all, 5 = I am always sure. The minimum score that can be obtained from the scale is 14, and the maximum is 70.
Mother to Infant Bonding Scale | 3 months
  Mother to Infant Bonding Scale is a measurement tool that can be applied from the first day after birth and allows the mother to express her feelings towards her baby in a single word.
  The lowest total score that can be obtained from the scale is 0 and the highest score is 24.
Father Breastfeeding Self-Efficacy Scale Short Form | 3 months
  This scale is a 14-item questionnaire that assesses a father's confidence in his ability to assist his partner with breastfeeding. The scale is in a 5-point Likert type and is evaluated as 1 = I am not sure at all, 5 = I am always sure. The minimum score that can be obtained from the scale is 14, and the maximum is 70.
Paternal -İnfant Attachment Questionnaire | 3 months
  The scale developed to evaluate postnatal father-infant attachment is a 19-item scale. Scale; It consists of three sub-dimensions: 'patience and tolerance', 'pleasure in interaction' and 'love and pride'. Each item of the scale is scored between 1 and 5 points. High scores indicate high attachment.
Baby Evaluation Form | 3 months
  The infant evaluation form was created by the researchers in line with the literature. In this form, there are questions about the height, weight and head circumference measurements of the babies, the way of feeding, whether they use pacifiers and bottles.

CONTACTS AND LOCATIONS:
Overall Officials: Ayfer Açıkgöz, Principal Investigator — ayferackgoz@gmail.com
Locations (1):
- Eskişehir Osmangazi Üniversitesi Sağlık Bilimleri Fakültesi, Eskişehir, Turkey (Türkiye)

REFERENCES:
- [Background] Abbass-Dick J, Dennis CL. Breast-feeding Coparenting Framework: A New Framework to Improve Breast-feeding Duration and Exclusivity. Fam Community Health. 2017 Jan/Mar;40(1):28-31. doi: 10.1097/FCH.0000000000000137. PMID 27870751
- [Background] Abbass-Dick J, Stern SB, Nelson LE, Watson W, Dennis CL. Coparenting breastfeeding support and exclusive breastfeeding: a randomized controlled trial. Pediatrics. 2015 Jan;135(1):102-10. doi: 10.1542/peds.2014-1416. Epub 2014 Dec 1. PMID 25452653
- [Background] Abbass-Dick J, Xie F, Koroluk J, Alcock Brillinger S, Huizinga J, Newport A, Goodman WM, Dennis CL. The Development and piloting of an eHealth breastfeeding resource targeting fathers and partners as co-parents. Midwifery. 2017 Jul;50:139-147. doi: 10.1016/j.midw.2017.04.004. Epub 2017 Apr 18. PMID 28448858
- [Background] Bennett AE, McCartney D, Kearney JM. Views of fathers in Ireland on the experience and challenges of having a breast-feeding partner. Midwifery. 2016 Sep;40:169-76. doi: 10.1016/j.midw.2016.07.004. Epub 2016 Jul 4. PMID 27450588
- [Background] Beyene AM, Liben ML, Arora A. Factors associated with the early termination of exclusive breastfeeding among mother-infant dyads in Samara-Logia, Northeastern Ethiopia. BMC Pediatr. 2019 Nov 11;19(1):428. doi: 10.1186/s12887-019-1803-1. PMID 31711461
- [Background] Brown A, Davies R. Fathers' experiences of supporting breastfeeding: challenges for breastfeeding promotion and education. Matern Child Nutr. 2014 Oct;10(4):510-26. doi: 10.1111/mcn.12129. Epub 2014 Apr 10. PMID 24720518
- [Background] Dennis CL. The breastfeeding self-efficacy scale: psychometric assessment of the short form. J Obstet Gynecol Neonatal Nurs. 2003 Nov-Dec;32(6):734-44. doi: 10.1177/0884217503258459. PMID 14649593
- [Background] Dennis CL, Faux S. Development and psychometric testing of the Breastfeeding Self-Efficacy Scale. Res Nurs Health. 1999 Oct;22(5):399-409. doi: 10.1002/(sici)1098-240x(199910)22:53.0.co;2-4. PMID 10520192
- [Background] Dennis CL, Brennenstuhl S, Abbass-Dick J. Measuring paternal breastfeeding self-efficacy: A psychometric evaluation of the Breastfeeding Self-Efficacy Scale-Short Form among fathers. Midwifery. 2018 Sep;64:17-22. doi: 10.1016/j.midw.2018.05.005. Epub 2018 May 15. PMID 29864577
- [Background] Ingram J, Johnson D. A feasibility study of an intervention to enhance family support for breast feeding in a deprived area in Bristol, UK. Midwifery. 2004 Dec;20(4):367-79. doi: 10.1016/j.midw.2004.04.003. PMID 15571885
- [Background] Jensen D, Wallace S, Kelsay P. LATCH: a breastfeeding charting system and documentation tool. J Obstet Gynecol Neonatal Nurs. 1994 Jan;23(1):27-32. doi: 10.1111/j.1552-6909.1994.tb01847.x. PMID 8176525
- [Background] Kucukoglu S, Sezer HK, Dennis CL. Validity and reliability of the Turkish version of the paternal breastfeeding self-efficacy scale - Short form for fathers. Midwifery. 2023 Jan;116:103513. doi: 10.1016/j.midw.2022.103513. Epub 2022 Oct 22. PMID 36323075
- [Background] Maycock B, Binns CW, Dhaliwal S, Tohotoa J, Hauck Y, Burns S, Howat P. Education and support for fathers improves breastfeeding rates: a randomized controlled trial. J Hum Lact. 2013 Nov;29(4):484-90. doi: 10.1177/0890334413484387. Epub 2013 Apr 19. PMID 23603573
- [Background] Ogbo FA, Akombi BJ, Ahmed KY, Rwabilimbo AG, Ogbo AO, Uwaibi NE, Ezeh OK, Agho KE, On Behalf Of The Global Maternal And Child Health Research Collaboration GloMACH. Breastfeeding in the Community-How Can Partners/Fathers Help? A Systematic Review. Int J Environ Res Public Health. 2020 Jan 8;17(2):413. doi: 10.3390/ijerph17020413. PMID 31936302
- [Background] Ozluses E, Celebioglu A. Educating fathers to improve breastfeeding rates and paternal-infant attachment. Indian Pediatr. 2014 Aug;51(8):654-7. doi: 10.1007/s13312-014-0471-3. PMID 25129001
- [Background] Pisacane A, Continisio GI, Aldinucci M, D'Amora S, Continisio P. A controlled trial of the father's role in breastfeeding promotion. Pediatrics. 2005 Oct;116(4):e494-8. doi: 10.1542/peds.2005-0479. PMID 16199676
- [Background] Rempel LA, Rempel JK, Moore KCJ. Relationships between types of father breastfeeding support and breastfeeding outcomes. Matern Child Nutr. 2017 Jul;13(3):e12337. doi: 10.1111/mcn.12337. Epub 2016 Jul 27. PMID 27460557
- [Background] Susin LR, Giugliani ER. Inclusion of fathers in an intervention to promote breastfeeding: impact on breastfeeding rates. J Hum Lact. 2008 Nov;24(4):386-92; quiz 451-3. doi: 10.1177/0890334408323545. Epub 2008 Sep 10. PMID 18784322
- [Background] Smith MM, Durkin M, Hinton VJ, Bellinger D, Kuhn L. Initiation of breastfeeding among mothers of very low birth weight infants. Pediatrics. 2003 Jun;111(6 Pt 1):1337-42. doi: 10.1542/peds.111.6.1337. PMID 12777550
- [Background] Su M, Ouyang YQ. Father's Role in Breastfeeding Promotion: Lessons from a Quasi-Experimental Trial in China. Breastfeed Med. 2016 Apr;11:144-9. doi: 10.1089/bfm.2015.0144. Epub 2016 Feb 2. PMID 26836960
- [Background] Taylor A, Atkins R, Kumar R, Adams D, Glover V. A new Mother-to-Infant Bonding Scale: links with early maternal mood. Arch Womens Ment Health. 2005 May;8(1):45-51. doi: 10.1007/s00737-005-0074-z. Epub 2005 May 4. PMID 15868385
- [Background] Wu W, Zhang J, Silva Zolezzi I, Fries LR, Zhao A. Factors influencing breastfeeding practices in China: A meta-aggregation of qualitative studies. Matern Child Nutr. 2021 Oct;17(4):e13251. doi: 10.1111/mcn.13251. Epub 2021 Aug 6. PMID 34355869
- [Background] Cakirli M, Acikgoz A. A Randomized Controlled Trial: The Effect of Own Mother's Breast Milk Odor and Another Mother's Breast Milk Odor on Pain Level of Newborn Infants. Breastfeed Med. 2021 Jan;16(1):75-81. doi: 10.1089/bfm.2020.0222. Epub 2020 Oct 20. PMID 33085532
- See also: Emzirme Tutumunu Değerlendirme Ölçeği — https://dergipark.org.tr/en/download/article-file/207494
- See also: Ebeveynlere Verilen Emzirme Eğitiminin Emzirme Öz-Yeterlilik Düzeyi Sadece Anne Sütü İle Beslenme Süresi ve Ebeveyn Bebek Bağlanmasına Etkisi — https://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp
- See also: Term Bebeklerde Ayak Topuğundan Kan Alma İşlemi Sırasında Dinletilen Beyaz Gürültünün, Elle Verilen Cenin Pozisyonunun Ve Her İki Uygulamanın Birlikte Yapılmasının Ağrıya Etkisi — https://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp
- See also: Yenidoğan Yoğun Bakım Ünitesinde Yatan Bebeklerde Kan Alma İşlemi Sırasında Uygulanan Kendi Anne Sütü Kokusunun Ve Farklı Annenin Sütünün Kokusunun Bebeklerin Ağrı Düzeylerine Etkisi — https://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp
- See also: Emzirmenin Başarılmasında Anahtar Faktör: Baba Desteğinin Sağlanması Ve Hemşirenin Rolleri. — https://dergipark.org.tr/en/download/article-file/626788
- See also: Anne-Bebek Bağlanma Ölçeğinin Türk Toplumuna Uyarlanmasi: Aydın Örneği — https://dergipark.org.tr/en/download/article-file/222161
- See also: Türkiye Nüfus ve Sağlık Araştırması (TNSA), 2018 — http://fs.hacettepe.edu.tr/hips/dosyalar/Ara%C5%9Ft%C4%B1rmalar%20-%20raporlar/2018%20TNSA/TNSA2018_ana_Rapor_compressed.pdf
- See also: World Health Organization. Infant And Young Child Feding — https://www.who.int/news-room/fact-sheets/detail/infant-and-young-child-feeding